CLINICAL TRIAL: NCT04971304
Title: An Exploratory Comparative Effectiveness Analysis of Granulocyte Colony Stimulating Factor Originator Products Versus Biosimilars in Real-world Practice
Brief Title: Comparative Effectiveness Analysis of Granulocyte Colony Stimulating Factor Originator Products Versus Biosimilars
Status: Completed | Type: Observational
Sponsor: Catherine M. Lockhart (Other)
Collaborators: Harvard Pilgrim Health Care (Other); HealthPartners Institute (Other)
Responsible Party: Sponsor-Investigator, Catherine M. Lockhart, Executive Director, Biologics & Biosimilars Collective Intelligence Consortium
Organization: Biologics & Biosimilars Collective Intelligence Consortium (Other)
Other Study IDs: BBCIC-GCSF-02
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Cancer, Breast; Cancer, Lung; Cancer of Colon; Cancer of Pancreas; Cancer, Ovarian; Lymphoma, Non-Hodgkin
Keywords: colony stimulating factor
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- G-CSF originator receipt: Patients receiving filgrastim (Neupogen) or pegfilgrastim (Neulasta) per Health Care Procedural Coding System (HCPCS) J-codes.
  Interventions: Drug: Receipt of granulocyte-colony stimulating factor
- G-CSF biosimilar receipt: Patients receiving filgrastim biosimilars (filgrastim-aafi, filgrastim-sndz, tbo-filgrastim) or pegfilgrastim biosimilars (pegfilgrastim-jmdb, pegfilgrastim-bmez, pegfilgrastim-cbqv) per Health Care Procedural Coding System (HCPCS) J-codes.
  Interventions: Drug: Receipt of granulocyte-colony stimulating factor

INTERVENTIONS:
Drug: Receipt of granulocyte-colony stimulating factor — Receipt of originator or biosimilar

SUMMARY:
This comparative effectiveness and descriptive retrospective cohort study will evaluate safety and effectiveness outcomes among commercially insured adults who received a granulocyte colony stimulating factor (G-CSF) biosimilar or originator product during the first cycle of clinical guideline-indicated intermediate or high febrile neutropenia risk chemotherapy.

DETAILED DESCRIPTION:
This comparative effectiveness and descriptive retrospective cohort study includes commercially insured adults enrolled in one of four health plans participating in the Biologics and Biosimilars Collective Intelligence Consortium (BBCIC) Distributed Research Network. The investigators included patients who received a granulocyte colony stimulating factor (G-CSF) biosimilar or originator product during the first cycle of clinical guideline-indicated intermediate or high febrile neutropenia risk chemotherapy. The investigators will collect patient demographics, cancer diagnosis, chemotherapy regimen, and patterns of G-CSF biosimilar and originator product use. The investigators will follow patients from first G-CSF exposure until up to six cycles of chemotherapy receipt, death, or insurance disenrollment. The primary effectiveness outcome is incidence of febrile neutropenia. Secondary outcomes include incidence of adverse events and trends in product use over time. The investigators will compare febrile neutropenia incidence between originator and biosimilar products using inverse probability weighting to control for confounding. Secondary analyses will examine 'as treated' outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 20 or older
* Diagnosis of lung, breast, colon, ovarian, pancreatic, testicular, cervical, uterine, or NHL cancer
* Beginning intermediate or high neutropenia risk chemotherapy

Exclusion Criteria:

* One inpatient or two outpatient cancer diagnoses at least 30 days apart in the 183 days prior to the Index Date for cancer different from enrolling cancer diagnosis
* Any of the following in 183 days prior to Index Date:
* Any chemotherapy or G-CSF product receipt
* 2< medical claims at least 30 days apart for a skilled nursing facility or hospice care
* 2< diagnoses/procedure codes at least 1 day apart for cancer-related radiotherapy, bone marrow or stem cell transplant, diagnosis of HIV/AIDS, severe hepatic disease, chronic kidney disease, or any non-oncology related neutropenia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung, breast, colon, ovarian, pancreatic, testicular, cervical, uterine, or NHL cancers initiating clinical guideline-indicated intermediate or high neutropenia risk chemotherapy between March 1, 2015 and December 31, 2019. Study period observation ends by June 30, 2020 for participant follow-up. A 12-month look-back prior to the study period (i.e. as early as March 1, 2014) will be used to ensure health plan enrollment, find incident cancer diagnoses, and provide a description of reference G-CSF utilization before biosimilar introduction to the US market.
Sampling Method: Non-Probability Sample
Enrollment: 16506 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients who develop febrile neutropenia | Within 30 days of receipt of first chemotherapy
  ICD-9 or ICD-10 codes for inpatient or outpatient visit indicating fever with infection per validated algorithms.

SECONDARY OUTCOMES:
Number of patients who develop G-CSF associated adverse events | Within 30 days of receipt of first chemotherapy
  ICD-9 or ICD-10 codes indicating splenic rupture, anaphylaxis, or leukocytosis.

IPD SHARING:
Plan to Share IPD: No